CLINICAL TRIAL: NCT02953470
Title: Community-dwelling Older Adults Living With Chronic Musculoskeletal Pain: The Effect of an Evidence-based Intervention on Pain, Function, Health and Behaviour
Brief Title: Effect Study of on Intervention on Pain, Function, Health and Behaviour for Older Adults Living With Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OsloAUCAS2016/859
Record Dates: First submitted 2016-10-21; First posted 2016-11-02 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; community-dwelling; older adults; physical activity; physiotherapy; behavioural medicine; biopsychosocial; exercise; independency; everyday activities; self-efficacy; quality of life; pain-related beliefs; pain-related disability
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual tailored functional exercise (Experimental): Receives general advice about physical activity with the goal to be physically active at least 30 minutes per day at 5 of 7 days per week. The intervention group, which is based on a behavioural medicine approach in physiotherapy, also receive individual tailored functional exercise with the goal to enhance the ability to perform everyday activities by reduce pain-related disability and pain-related beliefs and increase physical function. The participants receive 9 visits from a physiotherapist during the 12 weeks period. The participants will also fill in a activity diary to check the compliance to the intervention and to enhance their self-efficacy in relation to perform everyday activities, exercise and physical activity.
  Interventions: Behavioral: Individual tailored functional exercise
- Standard care (Active Comparator): The participants in the comparison Group will receive standard care which means that they receives one visit from physiotherapist where the participant receive general advice about physical activity with the goal to be physically active at least 30 minutes per day at 5 of 7 days per week. During intervention week 1-8 and 10 the participants receive telephone calls once a week where they will be reminded to follow the advice about physical activity.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Individual tailored functional exercise — Receive individual tailored exercise to increase ability to perform everyday activities through increased physical function and self-efficacy in relation to be able to exercise and decreased pain-related beliefs such as fear of falling, catastrophizing thoughts and fear of movement.
  Arms: Individual tailored functional exercise
Behavioral: Standard care — Receives written and oral advice about physical Activity and the benefits of being physically active by one visits from a physiotherapist. Than will the participants receive Telephone reminder about following the advice once a week during intervention week 1-8 and 10.
  Arms: Standard care

SUMMARY:
The aim for the study is to examined the effect of an individually tailored integrated behavioral medicine in physiotherapy intervention including functional exercise, for older adults, having chronic musculoskeletal pain, living alone and dependent on formal care.

The study is a pragmatic randomized controlled trial with one intervention group and one control group. The intervention is a 12-weeks home-based program. The intervention consists of an individually tailored intervention and aims to enhance ability to perform everyday activities by improving physical function and reduce pain-related beliefs and pain-related disability. The comparison group achieves general advice about physical activity. All participants will be tested at baseline, a post-assessment at 12 week and a three month follow-up. Primary outcome is pain interference by the Brief Pain Inventory and physical function by Short Physical Performance Battery.

Secondary outcomes measures if the goal setting is reached, self-efficacy in relation to the goal setting, pain catastrophizing, level of physical Activity, falls efficacy and Health related quality of life.

DETAILED DESCRIPTION:
Intervention group

The base for the intervention is to identify a problematic everyday activity and identify factors, including physical, psychological and environmental factors, that can inhibit and/or promote the ability to perform the activity. The exercise that will improve the physical factors will be based on functional exercise such as Balance training and muscle strength training, e.g. fast walking in circle, marching on the spot with a high knee lift, leg lifts, power walking and stair walking, squats, lunge, turning trunk and head while standing, and walking over obstacles. Number of exercises and the dosage are based on how much the participant are able to do and want to do and will increase progressively considering the changes in function and health status of the participants. The content of the visits is as follow:

Session: Identification of a problematic everyday activity and advice about physical activity.

Session 2: Doing functional behavioural analyse including goal setting, discuss performance dosage of training.

Session 3-5: Training in the basic physical and psychological skills relevant to goal setting.

Session 6-9: Training to apply basic skills adequately for the goal setting, application of basic and applied skills to other behaviours, starting with subsequent activity goals.

Discussion about how the participant can be able to maintain their new behaviour.

Discussion of problem-solving strategies, how he/she can prevent and address new activity problems that may arise related to the goal setting and in relation to being physically active.

During the intervention period will the participant receive visits by a physiotherapist during intervention weeks 1-8 and 12. Under week 10 will the participants receive one telephone call for support.

Non-intervention Group

The comparison group will receive standard care which means that the participants get one visit from physiotherapist which consist of written and oral information about general advice regarding physical Activity..Further will the comparison group receive telephone Calls to remind them of being physically active according to the advice during week 1-8 and week 10.

ELIGIBILITY:
Inclusion Criteria:

* 75 years, Living in the central part of Oslo, Norway Living alone in ordinary housing Dependent on home help services for individual care and/or housekeeping activities or home care for medical needs The presence of musculoskeletal pain for three month or longer Ability to walk independently indoors, with or without a walking aid Ability to understand and speak Norwegian Ability to fill in activity diary or to have someone to help them with that.

Exclusion Criteria:

Older adults ongoing physiotherapy treatment for injury/illness, Are in a palliative stage of treatment Have experienced heart failure in the past three months.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Pain-related disability measured with the pain interference score in Brief Pain Inventory (BPI) | six month
  Pain-related disability will be measured with the pain interference score in Brief Pain Inventory (BPI). The BPI is a self-report pain assessment tool and the patient is instructed to report pain as intensity and as interference with seven different functions. The interference scale includes seven items which assess pain's interference with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life. The BPI has shown to be The BPI is validated for use in older adults with non cancer pain.
Physical function measured by the Norwegian version of the Short Physical Performance Battery | six month
  Physical function will be measured by the Norwegian version of The short physical performance battery. The Short Physical Performance Battery (SPPB) evaluates balance, mobility and muscle strength by examining an individual's ability to stand with feet together in side-by side, semi-tandem and tandem positions, time to walk 8 ft and time to rise from a chair and return to the seated position five times. Each of the three tests is scored, based on performance between 0 and 4, leaving a maximum score of 12 for those individuals performing at the highest levels. The SPPB is a reliable and valid measure of lower extremity performance. Meaningful changes in the SPPB have been defined. Thus, the SPPB can be used as a standard measure of physical performance both for research and in clinical practice.

SECONDARY OUTCOMES:
Reach of goal setting | three month
  For the participants in the intervention group will the following be checked: If the goal setting is reached or not will be measured by an Yes/No question
Pain severity measured by the BPI short version | six month
  Pain severity measured by the BPI short version. The BPI is a self-report pain assessment tool and the patient is instructed to report pain as intensity and as interference with seven different functions (49). The intensity scale contains four items measuring worst, least and average pain intensity (usually during the past 24 hours or past week) and intensity now.
Pain catastrophizing measured by the Catastrophizing subscale | six month
  will be measured with two items from the Catastrophizing subscale which is a part of the Coping strategies questionnaire.
Falls efficacy measured by the Norwegian version of the Falls-Efficacy Scale international (FES-I) | six month
  is measured by the Norwegian version of the Falls-Efficacy Scale international (FES-I). The FES-I assesses level of concern about falling on a 4 point scale during 16 activities of daily living. Scores range from 16 to 64 with higher scores indicating greater concern about falling.
physical activity level according to a six-point scale | six month
  The level of physical activity, including housekeeping activities, was estimated for the summer and winter seasons according to a six-point scale. The scale ranged from "hardly any physical activity" (level 1) to "hard exercise several times a week" (level 6). The scale has been shown to be valid for older people.
Health related quality of life measured with SF-12 | six month
  will be measured with The Short Form Health survey,SF-12. SF-12 is a shortened version of SF-36 (55)) and has shown to be valid to use among older people.
Self-efficacy in relation to goal setting | three month
  The participants in the intervention Group will measure their self-efficacy in relation to the goal setting by and Self-efficacy in relation to the goal setting will be measured by a four-graded verbal descriptive scale; Not sure at all, little sure, rather sure, very sure.

OTHER OUTCOMES:
Consumer questions | at three and six month
  To assess the participants expected results of the intervention they will be asked to answer the following questions:
  How do you experience your physical activity level now after participation in the study? How do you experience your physical activity level now after participation in the study? 3) How are your physically problems now after ending the participation in the study? 4) Do you use what you learned during the intervention to manage or prevent your physically problem? 5) Describe how you use what you have learned to manage or prevent your physically problems 7) Do you take any pain medication more or less or the same Have you visit a physiotherapist Yes/no, if Yes, for what and what treatment did you get
Age | baseline
  Age (years)
Gender | baseline
  Gender; male/female
Home-help services | baseline
  Number of home help services
Home care | baseline
  Number of help from home care
Medical diagnoses | baseline
  self-reported number Medical diagnoses
Pain medication | baseline
  self-reported Number and use of pain medication
Years With pain | baseline
  Number of years With pain
Falls | baseline
  Number of falls last year
Physical activity | baseline
  If the participants are so physically active as they wish
Walking aid | baseline
  use of walking aid
Getting outdoors | baseline
  If get outdoors by them selves

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, Professor, Study Chair — Oslo Metropolitan University
Locations (1):
- Sara Cederbom, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cederbom, S. (2014). Ability in everyday activities and morale among older women with chronic musculoskeletal pain living alone. A behavioural medicine approach in physiotherapy (Doctoral Thesis), Karolinska Institutet, Stockholm,Sweden
- [Background] AGS Panel on Persistent Pain in Older Persons. The management of persistent pain in older persons. J Am Geriatr Soc. 2002 Jun;50(6 Suppl):S205-24. doi: 10.1046/j.1532-5415.50.6s.1.x. No abstract available. PMID 12067390
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Result] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Klepstad P, Loge JH, Borchgrevink PC, Mendoza TR, Cleeland CS, Kaasa S. The Norwegian brief pain inventory questionnaire: translation and validation in cancer pain patients. J Pain Symptom Manage. 2002 Nov;24(5):517-25. doi: 10.1016/s0885-3924(02)00526-2. PMID 12547051
- [Result] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Result] Helbostad JL, Taraldsen K, Granbo R, Yardley L, Todd CJ, Sletvold O. Validation of the Falls Efficacy Scale-International in fall-prone older persons. Age Ageing. 2010 Mar;39(2):259. doi: 10.1093/ageing/afp224. Epub 2009 Dec 22. No abstract available. PMID 20031925
- [Result] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Result] Jakobsson U, Westergren A, Lindskov S, Hagell P. Construct validity of the SF-12 in three different samples. J Eval Clin Pract. 2012 Jun;18(3):560-6. doi: 10.1111/j.1365-2753.2010.01623.x. Epub 2011 Jan 6. PMID 21210901
- [Result] Frändin K, Grimby G. Assessment of physical activity, fitness and performance in 76-year-olds. Scand J Med Sci Sports. 1994;4(1):41-6.
- [Result] Utne I, Miaskowski C, Bjordal K, Paul SM, Jakobsen G, Rustoen T. Differences in the use of pain coping strategies between oncology inpatients with mild vs. moderate to severe pain. J Pain Symptom Manage. 2009 Nov;38(5):717-26. doi: 10.1016/j.jpainsymman.2009.03.005. Epub 2009 Sep 22. PMID 19775862